CLINICAL TRIAL: NCT07247149
Title: Testing a Novel Attention Based Training Prevention Strategy for First Responders: FirstFocus a Mobile Appt
Brief Title: Testing a Novel Attention Based Training Prevention Strategy for First Responders: FirstFocus a Mobile App
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto University (Other)
Responsible Party: Principal Investigator, Mikael Rubin, Assistant Professor, Palo Alto University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-024-PAU
Record Dates: First submitted 2025-11-19; First posted 2025-11-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Wellbeing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Attention Training Baseline Start (Experimental): Participants in this arm will begin ABM at the start of the study.
  Interventions: Behavioral: Attention Bias Modification
- Attention Training Week 1 Start (Experimental): Participants in this arm will begin ABM 1 week after the start of the study.
  Interventions: Behavioral: Attention Bias Modification
- Attention Training Week 2 Start (Experimental): Participants in this arm will begin ABM 2 weeks after the start of the study.
  Interventions: Behavioral: Attention Bias Modification
- Attention Training Week 3 Start (Experimental): Participants in this arm will begin ABM 3 weeks after the start of the study.
  Interventions: Behavioral: Attention Bias Modification

INTERVENTIONS:
Behavioral: Attention Bias Modification — Attention training involves 80 training trials. The task uses words developed specifically for this study with fear words such as "crash" and "car" and neutral words such as "couch" and "can" that are balanced for length and frequency. Additionally, on every trial the location of the probe is the same as the location of the fear word. Participants press the button corresponding to the direction of the probe. The training takes approximately 5 minutes to complete.

SUMMARY:
First responders are frequently exposed to high-stress and traumatic events, putting them at increased risk for mental health challenges such as posttraumatic stress disorder, anxiety, and depression. Access to traditional mental health services is often hindered by stigma, time constraints, and a lack of tailored resources. Mobile app-based interventions offer a promising solution due to their accessibility and potential to address mental health proactively and in a time sensitive way. Attention training has emerged as a simple way to prevent distress and the emergence of future mental health concerns. The proposed research will test a mobile app: FirstFocus which will leverage targeted attention training to prevent stress/distress during shifts and enhance the wellbeing of rural first responders. The specific aims are to (1) test the feasibility and acceptability of FirstFocus as an intervention for rural first responders; (2) to test the short-term preventative efficacy of attention training on state stress/distress and its longer-term efficacy for improving professional quality of life and reducing symptoms of anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Employed as an Active First Responder
* iPhone mobile device
* Located in a rural part of the US

Exclusion Criteria:

- Works less than 20 hours/week on average

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire | From enrollment to the end of treatment at 8 weeks.
  The Client Satisfaction Questionnaire - 8 item version (CSQ-8; Nguyen et al., 1983) will assess participant satisfaction with the FirstFocus app at the 60-day assessment. The CSQ-8 yields a total score ranging from 8 to 32, with higher scores indicating greater satisfaction.

SECONDARY OUTCOMES:
Stress Reduction (visual analogue scale) | From enrollment to the end of treatment at 8 weeks.
  Current stress will be assessed using a Visual Analogue Scale for Stress, administered daily before and after each shift. Participants rate their stress on a 0-100 scale, where 0 = no stress and 100 = extreme stress. Higher scores indicate greater stress.
Professional Quality of Life | From enrollment to the end of treatment at 8 weeks
  The Professional Quality of Life Scale, Version 5 (ProQOL-5) assesses compassion satisfaction, burnout, and secondary traumatic stress. Each subscale yields a score from 10 to 50, with higher Compassion Satisfaction scores reflecting better outcomes, and higher Burnout or Secondary Traumatic Stress scores reflecting worse outcomes. Administered weekly on login.
Symptoms of depression | From enrollment to the end of treatment at 8 weeks
  The Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2001) assesses depressive symptoms over the past week. Total scores range from 0 to 27, with higher scores indicating more severe depressive symptoms. Administered monthly on login.
Symptoms of anxiety | From enrollment to the end of treatment at 8 weeks
  The Generalized Anxiety Disorder-7 (GAD-7; Spitzer et al., 2006) assesses anxiety symptoms over the past week. Total scores range from 0 to 21, with higher scores indicating more severe anxiety. Administered monthly on login.
Stress | From enrollment to the end of treatment at 8 weeks
  The Perceived Stress Scale - 10 item version (PSS-10; Cohen et al., 1983) assesses perceived stress over the past week. Total scores range from 0 to 40, with higher scores indicating higher perceived stress levels. Administered monthly on login.

OTHER OUTCOMES:
Qualitative Evaluation of Acceptability. | From enrollment to the end of treatment at 8 weeks
  Qualitative feedback will be collected via a single open-ended item each week, along with multiple open-ended acceptability questions at the 60-day assessment. As a qualitative measure, no numerical scale or score range applies. This approach allows for detailed feedback on usability, acceptability, and alignment with first responder needs.

CONTACTS AND LOCATIONS:
Locations (1):
- Palo Alto University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All deidentified outcomes will be shared at the time of publication.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD and supporting information will be available at the time of publication of related findings/outcomes.